CLINICAL TRIAL: NCT07161934
Title: A Randomized Controlled Trial on the Effects of Guided Imagery Training on Shooting Accuracy and Psychological Skills in Adolescent Football Players
Brief Title: Guided Imagery Training for Shooting Accuracy and Mental Skills in Adolescent Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Burcu Güler (Other)
Responsible Party: Sponsor-Investigator, Merve Burcu Güler, Lecturer, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMAGERY-FOOTBALL-2020; 350-50 (Other: Çağ University, Institute of Social Sciences Ethics Committee)
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Adolescent; Soccer Performance; Psychological Phenomena and Processes; Imagery, Psychotherapy
Keywords: Guided Imagery; Mental Training; Shooting Accuracy; Sport Imagery; Psychological Skills; Youth Athletes; Football (Soccer); Performance

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to either the intervention group or the control group. The intervention group received guided imagery training in addition to standard football practice, while the control group received standard football training only. Both groups trained in parallel over a 12-week period, with outcomes assessed before and after the intervention.
Masking Description: Since participants and providers were aware of group allocation, the study was conducted as open label. However, statistical analyses were performed by an independent researcher blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery Training (Experimental): Participants in this arm received guided imagery training in addition to their standard football practice. After each 60-minute technical training session, a 15-minute guided imagery session was conducted, three times per week for 12 weeks (36 sessions total). The program included relaxation, visualization of technical movements, and reinforcement of confidence and motivation.
  Interventions: Behavioral: Guided Imagery Training
- Standard Football Training (Active Comparator): Participants in this arm received only standard football training, three times per week for 12 weeks (36 sessions total). To balance contact time, they attended 15-minute team evaluation meetings after each training session, but no imagery training was provided.
  Interventions: Behavioral: Standard Football Training

INTERVENTIONS:
Behavioral: Guided Imagery Training — Participants received guided imagery sessions of 15 minutes after each football training, three times per week for 12 weeks (36 sessions). Sessions included relaxation, visualization of technical movements, and reinforcement of motivation and confidence.
  Other Names: Mental Imagery; Sport Imagery
  Arms: Guided Imagery Training
Behavioral: Standard Football Training — Participants received only regular football training three times per week for 12 weeks (36 sessions). Each session lasted 60 minutes and focused on technical skills. To match contact time, a 15-minute team evaluation meeting was held after each practice.
  Other Names: Technical Training Only
  Arms: Standard Football Training

SUMMARY:
This study is designed to examine whether guided imagery training can improve football shooting performance and psychological skills in young athletes. Thirty-two male players aged 12-14 years will be randomly assigned to an imagery training group or a control group. The imagery group will receive guided mental training sessions after each regular football practice for 12 weeks, while the control group will participate only in standard training. The primary outcome will be shooting accuracy at 10 and 15 meters, and the secondary outcome will be imagery ability assessed with a validated questionnaire.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to evaluate the effects of a structured guided imagery program on shooting accuracy and sport-specific psychological abilities in adolescent football players. A total of 32 licensed male players, aged between 12 and 14 years, will be recruited from a local sports club and randomly assigned to one of two groups.

The intervention group will receive guided imagery sessions of 15 minutes following each of their three weekly football practices, over a total period of 12 weeks (36 sessions). These sessions will include relaxation, visualization of technical movements, and reinforcement of confidence and motivation. The control group will continue with standard technical training and will participate in short team meetings to match the contact time.

The primary outcome will be shooting accuracy, evaluated with a standardized shooting accuracy test at distances of 10 and 15 meters. The secondary outcome will be imagery ability, measured using the Sport Imagery Questionnaire for Children (SIQ-C).

The study design is a single-center, parallel-group randomized controlled trial. Ethical approval was obtained from the Institute of Social Sciences Ethics Committee at Çağ University (Approval No. 350-50, January 10, 2020). All participants and their parents will provide written informed consent before the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescent football players
* Age between 12 and 14 years
* Licensed players of Yozgat Municipality Bozok Sports Club
* Regular attendance at training sessions
* Written informed consent obtained from both player and parent/guardian

Exclusion Criteria:

* Withdrawal of consent at any time
* Health problems arising during the intervention that prevent participation
* Irregular or insufficient attendance at training sessions
* Female athletes (not available in this age category at the club)

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Shooting Accuracy Test (10 m and 15 m) | Baseline and 12 weeks (post-intervention).
  Change in football shooting accuracy measured with a standardized Shooting Accuracy Test at baseline and after 12 weeks. Players performed 10 shots with their dominant foot at distances of 10 m and 15 m, and the number of successful hits was recorded. Higher values indicate better shooting accuracy.

SECONDARY OUTCOMES:
Sport Imagery Questionnaire for Children (SIQ-C) Total and Subscale Scores | Baseline and 12 weeks (post-intervention).
  Change in total score and subscales (Specific Cognitive-Motivational, General Cognitive, and General Motivational-Mastery) of the Sport Imagery Questionnaire for Children (SIQ-C), a validated 21-item self-report questionnaire assessing imagery ability in children and adolescents. Each item is rated on a Likert scale from 1 to 5, resulting in total scores ranging from 21 to 105. Higher scores indicate greater imagery ability.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Burcu Güler, MSc in Psychology, Principal Investigator — Selcuk University, Vocational School of Health Services; Ayşe Avcı, PhD, Study Director — Çağ University, Institute of Social Sciences; Hayrettin Gümüşdağ, PhD, Study Chair — Yozgat Bozok University, Faculty of Sport Sciences
Locations (1):
- Yozgat Municipality Bozok Sports Club, Yozgat, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available from the corresponding author upon reasonable request after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data will be available beginning 6 months after publication of the main results and will be accessible for 5 years.
Access Criteria: Data will be shared with qualified researchers for academic purposes. Requests should be directed to the corresponding author (Merve Burcu Güler) via email. Access will be granted after review and approval of a reasonable request, and data will be shared in electronic format.